CLINICAL TRIAL: NCT06761209
Title: Is Negativity of Autoantibodies a Marker of Severity in Auto-immune Hepatitis
Brief Title: Is Negativity of Autoantibodies a Marker of Severity in Auto-immune Hepatitis?
Acronym: HAI-NEG
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2020/21; 2020-A02908-31 (Other: ANSM)
Record Dates: First submitted 2024-12-18; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Auto-immune Hepatitis
Keywords: autoantibodies; auto-immune hepatitis; prognosis; afrocaribbean population
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- acute or chronic Auto-Immune Hepatitis patients: For the study, a blood sample will be collected from the patient in order to build up a serological library which allow the search for rare autoAb whose interest has been demonstrated as prognostic factors of the disease
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — For the study, a blood sample will be collected from the patient in order to do build up a serological library which will allow the search for rare autoAb whose interest has been demonstrated as prognostic factors of the disease.

SUMMARY:
Evaluate the proportion of seronegative auto-immune hepatitis and a possible relationship with the severity of the disease. Criteria of severity will be defined by corticodependance, corticoresistance and a severe form of the disease at diagnosis (cirrhosis or fulminant hepatitis). In case of predominant seronegative forms, other auto-antibodies related to this auto-immue hepatitis will be searched.

DETAILED DESCRIPTION:
Evaluate the proportion of seronegative auto-immune hepatitis and a possible relationship with the severity of the disease. Criteria of severity will be defined by corticodependance, corticoresistance and a severe form of the disease at diagnosis (cirrhosis or fulminant hepatitis). In case of predominant seronegative forms, other auto-antibodies related to this auto-immue hepatitis will be searched.

Patients from the Guadeloupean constitutive center of rare diseases (CCRD Filfoie) and from the Saint-Antoine hospital will be retrospectively analyzed, and new patients will be prospectively followed.

ELIGIBILITY:
Inclusion Criteria:

* - Any patient over 18 years old
* Patient followed at Hôpital Saint-Antoine or treated for HAI or in Guadeloupe within the framework of the CCRD Filfoie for an acute or chronic AIH under immunosuppressive treatment
* Patient affiliate or beneficiary of a social security scheme
* Free, informed and written consent signed by the patient and the investigator

  o exclusion criteria: - Patient under 18 years old
* Patient not able to give his/her consent
* Viral hepatitis: viruses A to E, Epstein-Barr virus, cytomegalovirus and herpes simplex virus
* Isolated primary biliary cholangitis
* Isolated primary sclerosing cholangitis
* Drug-induced liver injury
* Wilson disease
* Alcoholic hepatitis
* Hemochromatosis
* Sickle cell disease and heart liver
* Non-alcoholic steato-hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: only acute or chronic AIH patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
histological rereading of seronegative AIH | Baseline
  Percentage comparisons will be made by a chi-2 test or a Fischer test.

SECONDARY OUTCOMES:
assessment of the severity of the disease | 6 months, 12 months
  - Number of corticosteroid HAI defined by the maintenance of corticosteroid therapy> 20mg / d beyond 6 months of treatment - Number of corticosteroid-resistant AIH. Percentage comparisons will be made by a chi-2 test or a Fischer test.
Constitution of a serotheque in order to search for other autoAb described as correlated to the severity of the AIH. | At inclusion
  Constitution of a serotheque in order to search for other autoAb described as correlated to the severity of the AIH.

CONTACTS AND LOCATIONS:
Overall Officials: Moana Lemoinne, doctor, Principal Investigator — chu de pointe à pitre
Locations (2):
- France (2):
  - Hospital of Saint-Antoine, Paris, France
  - CHU de Pointe-à Pitre, Pointe à Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No